CLINICAL TRIAL: NCT06014242
Title: Peripheral Microvascular Resistance as a Predictor for Limb Salvage in Post-Intervention Critical Limb Ischemia Patients
Brief Title: Peripheral Microvascular Resistance as a Predictor for Limb Salvage
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never opened to enrollment
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro2021-0681
Record Dates: First submitted 2023-08-21; First posted 2023-08-28 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Arterial Disease
Keywords: Microvascular disease; Microvascular Resistance; Limb Salvage; Peripheral Arterial Disease; critical limb ischemia
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Peripheral vascular flow reserve measurement (Experimental): Post-procedure peripheral vascular flow reserve by thermodilution will be measured by the pressure wire.
  Interventions: Diagnostic Test: Peripheral vascular flow reserve measurement

INTERVENTIONS:
Diagnostic Test: Peripheral vascular flow reserve measurement — Peripheral arterial (below knee popliteal and above the level of ankle distal tibial) thermodilution curves will be obtained. One of the distal tibial arteries (anterior tibial, posterior tibial or peroneal artery, whichever reaches the most distal part of the foot in the run off) will be picked for measurements. At room temperature, 3 ml of saline will be injected brisk manually to determine the peak arterial flow, presented as mean transit time (Tmn). Resting Tmn will be performed and averaged by triplicate measurements at baseline. Then maximal hyperemia will be induced by intra-arterial injection of 30 mg papaverine through the guiding catheter, then 3 ml of saline will be injected to get hyperemic Tmn averaged by triplicate measurements. The guidewire will be kept in a fixed position during the series of measurements. Peripheral vascular flow reserve was calculated as resting Tmn divided by hyperemic Tmn (Fukunaga 2015).

SUMMARY:
Salvaging a threatened limb is the key therapeutic objective for patients with critical limb ischemia, and the achievement of limb salvage is an independent predictor of patient morbidity and mortality. Despite successful primary endovascular or surgical intervention, the corresponding symptoms of rest pain and/or non-healing ulceration in some patients may continue, and amputation in these patients is unavoidable. It is hypothesized that the functional integrity of the peripheral vascular microcirculation may be impaired in these patients. However, there are currently no techniques that allow direct quantification and visualization of the microcirculation due to the micro-vessel invisibility under angiography.

In the coronary circulation, coronary flow reserve (CFR) indicates the capacity for maximal hyperemic blood flow and reveals impaired coronary microvascular function. Studies have shown the clinical significance of measuring microvascular resistance to predict myocardial salvage after myocardial infarction. The study will explore whether this concept of coronary flow reserve can be applied peripherally to patients with critical limb ischemia in order to determine whether measuring peripheral vascular flow reserve can determine the integrity of the microcirculation to predict limb salvage after endovascular intervention.

ELIGIBILITY:
Inclusion Criteria:

* Chronic critical limb ischemia (Rutherford 4-6).
* Age ≥18 years
* Ability and willingness to sign the IRB approved Informed Consent form

Exclusion Criteria:

* Non-reconstructable chronic total occlusive disease of the proximal inflow vessels that would make flow reserve measurements impossible.
* Non-salvageable lower extremity due to infection or overwhelming per-existing tissue loss (most critical Rutherford 6 patients).
* Inability to understand the study or a history of non-compliance with medical advice;
* History of any cognitive or mental health status that would interfere with study participation;
* Currently enrolled in any pre-approval investigational study.
* Female subjects who are pregnant or nursing or planning to become pregnant within the study period;
* Known sensitivity to contrast media, which can't be adequately pre-medicated;
* Expected life span less than 6 months.
* Unable to read/understand/sign the English Language consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the peripheral flow reserve | 6 months post-endovascular intervention
  To assess whether peripheral flow reserve can predict the success rate of limb salvage in critical limb ischemia patients after endovascular intervention. Assessed by any amputation (major or minor) at 6 months post-endovascular intervention.

SECONDARY OUTCOMES:
Symptom resolution - Ulcer healing (1m) | 1 month post-endovascular intervention
  Ulcer healing: changes in the number and extent of leg ulcers compared to baseline.
Symptom resolution - Ulcer healing (6m) | 6 months post-endovascular intervention
  Ulcer healing: changes in the number and extent of leg ulcers compared to baseline.
Number of patients with Symptom resolution - Pain (1m) | 1 month post-endovascular intervention
  Resolution of rest pain and alteration in visual analogue pain compared to baseline.
Number of patients with Symptom resolution - Pain (6m) | 6 months post-endovascular intervention
  Resolution of rest pain and alteration in visual analogue pain compared to baseline.
Ankle-brachial index (ABI) (1m) | 1 month post-endovascular intervention
  Improvement in Ankle-brachial index (ABI) compared to baseline. The Ankle Brachial Index (ABI) is the systolic pressure at the ankle, divided by the systolic pressure at the arm. Normal ABI ranges from 1.0 - 1.4, with <0.9 suggesting arterial disease.
Ankle-brachial index (ABI) (6m) | 6 months post-endovascular intervention
  Improvement in Ankle-brachial index (ABI) compared to baseline. The Ankle Brachial Index (ABI) is the systolic pressure at the ankle, divided by the systolic pressure at the arm. Normal ABI ranges from 1.0 - 1.4, with <0.9 suggesting arterial disease.
Toe-brachial index (TBI) (1m) | 1 month post-endovascular intervention
  Improvement in Toe-brachial index (TBI) compared to baseline. The Toe Brachial Index (TBI) is defined as the ratio between the systolic blood pressure in the right or left toe and the higher of the systolic pressure in the right or left arms. TBI ≥ 0.7 is considered normal while TBI < 0.7 is considered abnormal.
Toe-brachial index (TBI) (6m) | 6 months post-endovascular intervention
  Improvement in Toe-brachial index (TBI) compared to baseline. The Toe Brachial Index (TBI) is defined as the ratio between the systolic blood pressure in the right or left toe and the higher of the systolic pressure in the right or left arms. TBI ≥ 0.7 is considered normal while TBI < 0.7 is considered abnormal.
Rutherford classification (1m) | 1 month post-endovascular intervention
  Use of The Rutherford classification to assess peripheral artery disease compared to baseline. A 7 category scale is being used with 0 being Asymptomatic and 6 being Ulceration or gangrene.
Rutherford classification (6m) | 6 months post-endovascular intervention
  Use of The Rutherford classification to assess peripheral artery disease compared to baseline. A 7 category scale is being used with 0 being Asymptomatic and 6 being Ulceration or gangrene.
Transcutaneous oxygen partial pressure (TcPO2) (1m) | 1 month post-endovascular intervention
  Transcutaneous partial pressure of oxygen (TcPO2) will be measured representing the amount of oxygen diffusing outward across the skin (used as a surrogate for arterial perfusion).
Transcutaneous oxygen partial pressure (TcPO2) (6m) | 6 months post-endovascular intervention
  Transcutaneous partial pressure of oxygen (TcPO2) will be measured representing the amount of oxygen diffusing outward across the skin (used as a surrogate for arterial perfusion).
Target lesion revascularization (1m) | At 1 month post-endovascular intervention
  Need for revascularization (yes/no)
Target lesion revascularization (6m) | At 6 month post-endovascular intervention
  Need for revascularization (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: David O'Connor, MD, Principal Investigator — Hackensack Meridian Health

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGinn, A.L., White, C.W. and Wilson, R.F., 1990. Interstudy variability of coronary flow reserve. Influence of heart rate, arterial pressure, and ventricular preload. Circulation, 81(4), pp.1319-1330. Nahser Jr, P.J., Brown, R.E., Oskarsson, H., Winniford, M.D. and Rossen, J.D., 1995. Maximal coronary flow reserve and metabolic coronary vasodilation in patients with diabetes mellitus. Circulation, 91(3), pp.635-640. Payne, A.R., Berry, C., Doolin, O., McEntegart, M., Petrie, M.C., Lindsay, M.M., Hood, S., Carrick, D., Tzemos, N., Weale, P. and McComb, C., 2012. Microvascular resistance predicts myocardial salvage and infarct characteristics in ST-elevation myocardial infarction. Journal of the American Heart Association, 1(4), p.e002246. Camici, P.G., d'Amati, G. and Rimoldi, O., 2015. Coronary microvascular dysfunction: mechanisms and functional assessment. Nature Reviews Cardiology, 12(1), p.48.
- [Background] Fukunaga M, Fujii K, Kawasaki D, Nishimura M, Horimatsu T, Saita T, Miki K, Tamaru H, Imanaka T, Naito Y, Masuyama T. Vascular flow reserve immediately after infrapopliteal intervention as a predictor of wound healing in patients with foot tissue loss. Circ Cardiovasc Interv. 2015 Jun;8(6):e002412. doi: 10.1161/CIRCINTERVENTIONS.115.002412. PMID 26019143
- [Background] Crea, F., Lanza, G.A. and Camici, P.G., 2014. Mechanisms of coronary microvascular dysfunction. In Coronary Microvascular Dysfunction (pp. 31-47). Springer, Milano.
- [Background] Pijls NH, De Bruyne B, Smith L, Aarnoudse W, Barbato E, Bartunek J, Bech GJ, Van De Vosse F. Coronary thermodilution to assess flow reserve: validation in humans. Circulation. 2002 May 28;105(21):2482-6. doi: 10.1161/01.cir.0000017199.09457.3d. PMID 12034653
- [Background] Kern MJ. Coronary physiology revisited : practical insights from the cardiac catheterization laboratory. Circulation. 2000 Mar 21;101(11):1344-51. doi: 10.1161/01.cir.101.11.1344. PMID 10725297